CLINICAL TRIAL: NCT03606707
Title: Efficacy of Fluoroscopic Guided Atlantoaxial Joint Injection on Head and Neck Pain and Sleep Quality in RA Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, principle investigaror, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Atlantoaxial injection in RA
Record Dates: First submitted 2018-07-04; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Pain, Head; Sleep Disturbance
MeSH Terms: conditions — Headache; Parasomnias | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- corticosteroid (Experimental): steroid group, received intra-articular steroid injection for atlantoaxial joint. , in addition to methotrexate and chloroquine 400 mg per day.
  Interventions: Drug: Steroids
- oral steroid (No Intervention): systemic group, received systemic steroid 20 mg/d , in addition to methotrexate and chloroquine 400 mg per day.

INTERVENTIONS:
Drug: Steroids — intra-articular steroid injection for atlantoaxial joint
  Other Names: cortecosteroid
  Arms: corticosteroid

SUMMARY:
Efficacy of intra-articular steroid injection for inflamed atlantoaxial joint in patients with rheumatoid arthritis Inclusion criteria Patients with rheumatoid arthritis with MRI findings of atlantoaxial joint inflammation and failure of resolution after 2 weeks systemic steroid administration Exclusion criteria Coagulopathy, allergy to contrast material, pregnancy Interventional group (AS) group, received intra-articular steroid injection for atlantoaxial joint. , in addition to methotrexate and chloroquine 400 mg per day.

DETAILED DESCRIPTION:
Efficacy of intra-articular steroid injection for inflamed atlantoaxial joint on sleep quality and head and neck pain in patients with rheumatoid arthritis Inclusion criteria Patients with rheumatoid arthritis with MRI findings of atlantoaxial joint inflammation and failure of resolution after 2 weeks systemic steroid administration Interventional group (AS) group, received intra-articular steroid injection for atlantoaxial joint. , in addition to methotrexate and chloroquine 400 mg per day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis with MRI findings of atlantoaxial joint inflammation and failure of resolution after 2 weeks systemic steroid administration

Exclusion Criteria:

* Coagulopathy, allergy to contrast material, pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
neck pain | 3 months
  Visual analog scale 0-10

SECONDARY OUTCOMES:
neck disability | 3 months
  Oswestry Neck Pain Questionnaire 0-50
sleep quality | 3 months
  Pittsburgh sleep quality index

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hassanien, MD, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Manal Hassanien, Asyut, Assuit
  - Assiut governorate, Asyut

IPD SHARING:
Plan to Share IPD: Yes
Efficacy of intra-articular steroid injection for inflamed atlantoaxial joint in patients with rheumatoid arthritis Inclusion criteria Patients with rheumatoid arthritis with MRI findings of atlantoaxial joint inflammation and failure of resolution after 2 weeks systemic steroid administration Exclusion criteria Coagulopathy, allergy to contrast material, pregnancy Interventional group (AS) group, received intra-articular steroid injection for atlantoaxial joint. , in addition to methotrexate and chloroquine 400 mg per day.
Supporting Information: Study Protocol
Time Frame: 3 months